CLINICAL TRIAL: NCT04100122
Title: Luminex-based Assay to Identify Major IgE-binding Episode Among IgE-mediated Wheat-allergic Patient
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Samitivej Hospital group (Unknown)
Responsible Party: Sponsor
Other Study IDs: 359/2562(EC3)
Record Dates: First submitted 2019-09-17; First posted 2019-09-24 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Wheat Allergy
Keywords: Major allergen
MeSH Terms: conditions — Wheat Hypersensitivity | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum or plasma (Blood drawn will be done using 15 cc of blood volume)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Wheat-allergic: The diagnosis of IgE-mediated wheat allergy was made if they have one of the following criteria
  1. a convincing clinical history of the reactions within 4 hours after wheat ingestion during the past 12 months combined with positive skin prick test (SPT) and/or the level of specific IgE (sIgE) to wheat or
  2. a positive oral food challenge (OFC) result to wheat during the past 12 months
  Interventions: Procedure: Blood drawing
- Wheat tolerant: Patients with wheat tolerant confirmed by negative oral food challenge (OFC) result to wheat during the past 12 months
  Interventions: Procedure: Blood drawing
- Wheat oral immunotherapy: Patients with IgE-mediated wheat allergy and underwent wheat oral immunotherapy for at least 6 months or at the maintenance phase of the treatment
  Interventions: Procedure: Blood drawing

INTERVENTIONS:
Procedure: Blood drawing — Blood drawn will be done once using 15 mL of blood volume (Serum or plasma samples will be collected during the routine follow up of level of sIgE to wheat or during the oral food challenge test which intravenous insertion routinely prepared in case of the emergency reaction occurred). The specimen will be transferred to the Icahn School of Medicine at Mount Sinai, New York, USA for Laboratory processing (Luminex-based peptide assay)

SUMMARY:
This study will be using Luminex-based peptide assay (LPA) to determine major IgE-binding epitope among wheat allergic children to differentiate clinical phenotype.

DETAILED DESCRIPTION:
Luminex-based peptide assay (LPA) is a novel tool using machine learning techniques, developed to predict different degrees of food allergy has been successfully reported among cow's milk protein allergy. This technique provide a more precise and advanced adaptation from microarray-based immunoassay (MIA). Using this technique will aid us for the differentiation of clinical phenotypes of wheat-allergic patients. This study will be the first study to date using this technique aim to determine major IgE-binding epitope among immediated-reaction of wheat allergic children to differentiate clinical phenotypes, and may lead to further study to develop the new therapeutic approach to wheat-allergic patients.

ELIGIBILITY:
Inclusion criteria

1. Patients with IgE-mediated wheat allergy, with one of the following criteria; 1.1 a convincing clinical history of the reactions within 4 hours after wheat ingestion during the past 12 months combined with positive skin prick test (SPT) and/or the level of specific IgE (sIgE) to wheat or 1.2 a positive oral food challenge (OFC) result to wheat during the past 12 months OR
2. Patients with wheat tolerant confirmed by negative oral food challenge (OFC) result to wheat during the past 12 months OR
3. Patients with IgE-mediated wheat allergy and underwent wheat oral immunotherapy for at least 6 months or at the maintenance phase of the treatment

Exclusion criteria Patients with delayed allergic reactions after wheat ingestion greater than 4 hours

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients between the aged of 1-18 years with confirmed IgE-mediated wheat allergy will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Major Immunoglobulin (Ig) E-binding epitope on wheat proteins and serum/plasma of patients | 48 months
  For Luminex data, the binding intensity of antibody to epitope specific beads was calculated from the florescence signal of each bead. An index score of binding intensity was generated from the log2 transformation of the signal-to-background ratio and each peptide element, which was close to a normal distribution. A plate effect was observed and adjusted for using linear models. Antibody binding intensities (Luminex) from different groups were compared. To assess the changes in epitope-binding profiles, a linear model was used with group as a factor. Comparisons of interests were tested using t tests and resultant P-values were adjusted for multiple hypotheses using the Benjamini-Hochberg approach, which controls the false discovery rate (FDR) across epitopes. Epitopes were defined as differentially binding epitopes (DBE) if the FDR < 0.05 and fold changes (FCH) > 1.5.

SECONDARY OUTCOMES:
Predict different severity of wheat hypersensitivity reaction | 48 months
  For Luminex data, the binding intensity of antibody to epitope specific beads was calculated from the florescence signal of each bead. An index score of binding intensity was generated from the log2 transformation of the signal-to-background ratio and each peptide element, which was close to a normal distribution. A plate effect was observed and adjusted for using linear models. Antibody binding intensities (Luminex) from different groups were compared. To assess the changes in epitope-binding profiles, a linear model was used with group as a factor. Comparisons of interests were tested using t tests and resultant P-values were adjusted for multiple hypotheses using the Benjamini-Hochberg approach, which controls the false discovery rate (FDR) across epitopes. Epitopes were defined as differentially binding epitopes (DBE) if the FDR < 0.05 and fold changes (FCH) > 1.5.

CONTACTS AND LOCATIONS:
Overall Officials: witchaya srisuwatchari, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Suarez-Farinas M, Suprun M, Chang HL, Gimenez G, Grishina G, Getts R, Nadeau K, Wood RA, Sampson HA. Predicting development of sustained unresponsiveness to milk oral immunotherapy using epitope-specific antibody binding profiles. J Allergy Clin Immunol. 2019 Mar;143(3):1038-1046. doi: 10.1016/j.jaci.2018.10.028. Epub 2018 Dec 7. PMID 30528770